CLINICAL TRIAL: NCT02224131
Title: Randomized Comparison of Platelet Function Monitoring to Adjust Antiplatelet Therapy Versus a Common Antiplatelet Treatment for Intracranial Aneurysm Stent-assisted Coiling
Brief Title: Study of Antiplatelet Therapy for Intracranial Aneurysm Stent-assisted Coiling
Acronym: ATIASC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Youxiang Li, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT-1401
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Embolic Stroke
Keywords: platelet function test; stent;
MeSH Terms: conditions — Embolic Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monitoring Arm (Experimental): dose adjustment of both aspirin and clopidogrel in suboptimal responders identified based on a point of care assay(TEG)
  Interventions: Drug: Aspirin and clopidogrel
- Conventional Arm (Active Comparator): fixed dose regiment of both aspirin and clopidogrel in all patients following stent deployment according to international guidelines
  Interventions: Drug: Aspirin and clopidogrel

INTERVENTIONS:
Drug: Aspirin and clopidogrel — modification of aspirin and clopidogrelmaintenance doses based on a biological assay Device:thrombelastography(TEG) point of care assay TEG(Haemoscope Corporation, Niles, IL)
  Other Names: Aspirin Enteric Coated Tablets ,Bayer HealthCare AG ;; Plavix
Drug: Aspirin and clopidogrel — aspirin and clopidogrel maintenance doses (according to international guidelines)
  Other Names: Aspirin Enteric Coated Tablets; Plavix

SUMMARY:
Patients' responses to oral antiplatelet therapy are subject to variation. Bedside monitoring offers the opportunity to improve outcomes of intracranial aneurysm patients undergoing stent deployment by individualizing therapy.This trial is designed to demonstrate the superiority of a strategy of platelet function monitoring with dose adjustment in suboptimal responders as compared to a more conventional strategy without monitoring and without dose adjustment to reduce the primary end point evaluated 6 months after stent deployment in patients with intracranial aneurysms.

DETAILED DESCRIPTION:
Participating Centers : 10 China high neurointervention volume (>200) centers Rationale: Clopidogrel (75 mg/day), in combination with aspirin (100 mg/day), is currently the antiplatelet treatment of choice for prevention of stent thrombosis, and clinical trials have shown that, in high-risk patients, prolonged dual antiplatelet treatment is more effective than aspirin alone in preventing major thromboembolic events. However, despite the use of clopidogrel, a considerable number of patients continue to have thromboembolic events. Numerous in VITRO studies have shown that individual responsiveness to clopidogrel but also to aspirin is not uniform in all patients and is subject to inter- and intraindividual variability. The recent possibility of bedside monitoring of oral antiplatelet therapy offers the unique opportunity of tailoring antiplatelet therapy. However, the relevance of such strategy has never been evaluated in a randomized prospective adequately powered study of intracranial aneurysm patients. Late state stent thrombosis and after interruption of OAT, is another important safety issue raising the questions of the modalities of interruption of dual OAT within six months according to the most recent updated recommendations. When is the best interruption of dual OAT? Our first hypothesis is that a strategy of dose adjustment of OAT based on biological monitoring reduces the rate of the combined ischemic endpoints of death, stent thrombosis and stroke as compared to a conventional strategy (local practice without monitoring) in patients scheduled for intracranial stent implantation and followed up for six months. Our second hypothesis is that interruption of clopidogrel after 1.5 months of dual OAT is associated with a higher rate of the same combined ischemic endpoints as compared with patients in whom dual OAT is maintained for 3 months follow-up.

Objectives: 1) To demonstrate the superiority of the strategy of monitoring with dose adjustment in suboptimal responders (Monitoring Arm) as compared to a more conventional strategy (Conventional Arm) with fixed dose regimen of both oral antiplatelet agents in all patients as defined by the international guidelines to reduce the primary endpoint evaluated one year after DES implantation. 2) to demonstrate the superiority of a strategy of pursuit of a dual OAT beyond 3 months(Pursuit Arm) as compared to a strategy of interruption for 1.5 months(Interruption Arm).

Duration of the participation : from 18 up to 30 months according to the time delay from study start to randomization. No participants will be excluded from the study at the exception of consent withdrawal. However, participants who have not been randomized for interruption or continuation of DAPT at the 6 month follow up visit will terminate the study

Number of patients: 1856 patients. This number was obtained for the demonstration of the superiority of the strategy of monitoring (Monitoring Arm) over the conventional strategy (Conventional Arm) to reduce the primary endpoint by 33% (relative risk reduction).

Expected results: The ARCTIC study will provide answers to two major clinical challenges. It will also give a unique opportunity to assess the prevalence and the associated risk factors of suboptimal answers to OAT, but also to improve a suboptimal biological response. Finally, the economic impact of both strategies of monitoring and of interruption will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years) in whom elective intracranial stent placement is scheduled after diagnostic angiography
* Patients not treated by GPIIb/IIIa inhibitors prior to randomization.
* Provided written consent for participation in the trial prior to any study-specific procedures or requirements

Exclusion Criteria:

* •Oral anticoagulation (Vitamin K Antagonists).

  * Contraindication for aspirin and/or clopidogrel or GPIIb/IIIa inhibitors or to increasing dose of clopidogrel or aspirin
  * Ongoing or recent bleeding and/or recent major surgery (<3 weeks)
  * Severe liver dysfunction
  * Thrombocytopenia (Platelet count <80000/µl).
  * IIb/IIIa inhibitors within a week prior to randomization
  * multiple intracranial aneurysms
  * Patient at risk of poor compliance to the study
  * Patient not affiliated to social security
  * Pregnant women, no signed inform consent
  * Any invasive or surgical planned intervention during the year after stent placement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1856 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
ischemia stroke | within 6 months after the stent placement
  Evidence of clinically definite ischemic stroke confirmed by MRI

SECONDARY OUTCOMES:
bleeding | within 6 months after stent placement
  Evidence of clinically definite bleeding complication confirmed by CT or clinical symptoms

OTHER OUTCOMES:
recurrence of aneurysm, all causes of death | within 6 months after stent placement
  Evidence of clinically definite recurrence of aneurysm confirmed by DSA

CONTACTS AND LOCATIONS:
Overall Officials: Youxiang Li, Professor, Study Chair — Department of neurointervention of Beijing Neurosurgical Institute,capital medical university ,China
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Collet JP, Cuisset T, Range G, Cayla G, Elhadad S, Pouillot C, Henry P, Motreff P, Carrie D, Boueri Z, Belle L, Van Belle E, Rousseau H, Aubry P, Monsegu J, Sabouret P, O'Connor SA, Abtan J, Kerneis M, Saint-Etienne C, Barthelemy O, Beygui F, Silvain J, Vicaut E, Montalescot G; ARCTIC Investigators. Bedside monitoring to adjust antiplatelet therapy for coronary stenting. N Engl J Med. 2012 Nov 29;367(22):2100-9. doi: 10.1056/NEJMoa1209979. Epub 2012 Nov 4. PMID 23121439